CLINICAL TRIAL: NCT04598152
Title: Modulating Default Mode Network Function: A Transcranial Direct Current Stimulation (TDCS) Pilot Study
Acronym: MDMN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid restrictions prevented continuation during the funding window
Sponsor: Jay Fournier (Other)
Responsible Party: Sponsor-Investigator, Jay Fournier, Assistant Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY19090112
Record Dates: First submitted 2020-10-10; First posted 2020-10-22 (Actual); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The first part of the study consists of screening procedures that are meant to determine if potential participants are eligible to take part in the remainder of the study.
  If you qualify to take part in the scanning portion of the study, you will have 2 scanning sessions on separate days approximately a week apart. For each scan session you will undergo a functional Magnetic Resonance Imaging (fMRI) scan that lasts approximately 30 minutes and no more than 1 hour. The total time you will spend for each scan session will be between 1-3 hours.
  During the scanning session you will receive transcranial direct current stimulation (tDCS). Prior to scanning, sponge-electrodes will be placed on your scalp. These electrodes will be connected to a stimulator. This stimulator will apply weak currents to the brain while the MRI takes pictures of your brain's responses. The stimulation current that you will experience is usually less than a 6-volt battery but may be increased up to 15-volts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcranial Direct Current Stimulation during fMRI (Experimental): Each subject will undergo transcranial direct current stimulation twice while completing a task in the functional magnetic resonance imaging scanner.
  Interventions: Device: TDCS - transcranial direct current stimulation

INTERVENTIONS:
Device: TDCS - transcranial direct current stimulation — TDCS involves passing a weak current through the brain. One variant, cathodal TDCS, can be used to temporarily hyperpolarize cortical pyramidal cells, thereby decreasing neuronal connections. TDCS has been explored as a possible treatment for depression, but results to date are mixed. No work has examined whether TDCS can be used in an individually guided manner to target locations in the parietal cortex and alter the patterns of circuitry dysfunction described previously.

SUMMARY:
The primary purpose of this research is to gather scientific information about how different people's brains work when they look at different types of pictures. This will help to improve the investigators' understanding of the way the brain works for people who are depressed or anxious, and this knowledge could help lead to better diagnosis and treatment.

DETAILED DESCRIPTION:
In this study the investigators are examining the effects of weak electrical stimulation on brain activity as measured by functional magnetic resonance imaging (fMRI). MRI is a widely used method to obtain high resolution brain pictures that are routinely used for diagnostic and clinical purposes. The electrical stimulation is applied on the scalp with a non-FDA approved method called tDCS (transcranial Direct Current Stimulation), typically equivalent to what a 6V battery would produce (and up to no more than 15V). To compare, an AA battery delivers current at 1.5 volt. While almost unnoticeable to the participants, these currents can still temporarily affect brain activity without causing adverse effects. This stimulation would be applied while the participants are in the MRI scanner so that the brain activity can be measured. The participants will have the opportunity to have a test session with the stimulation outside the scanner to get familiar with it.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-30years old
2. Score > 10 on the QIDS or > 60 on the PROMIS-A
3. We will use a flexible extreme groups recruitment strategy to ensure an adequate distribution of ESC scores. We will ensure that at least 62% of the sample will be composed of those scoring .5 SD above or below the mean, as measured by the NEO-PI-R. This value corresponds to the expected values assuming a normal distribution of the trait.
4. Normal or corrected to normal vision with contact lenses
5. Able to provide informed consent in English
6. Right-handed (Annett criteria)

Exclusion Criteria:

1. Have a history of head trauma with loss of consciousness.
2. Have a systemic medical illness that may impact fMRI measures of cerebral blood flow.
3. Meet standard exclusion criteria for fMRI scanning (e.g. claustrophobia, cardiac pacemakers, neural pacemakers, surgically implanted metal devices, cochlear implants, metal braces, or other MRI non-safe metal objects in the body).
4. Are pregnant (self report and tested for as part of any scan by the scanning center and not this protocol)
5. Not native English speaking or not fluent
6. Premorbid NAART IQ estimate<85;
7. Visual disturbance (worse than 20/40 Snellen visual acuity) that is not corrected
8. If have visual disturbance, only access to correction with glasses (i.e., no access to contact lenses).
9. Left/mixed handedness (Annett criteria), to ensure a uniform hemispheric dominance for interpretation of neuroimaging data
10. Active suicidal ideation in need of immediate treatment
11. Scoring below the cutoffs on both the QIDS and the PROMIS-A
12. History of alcohol/substance use disorder (including nicotine) and/or illicit substance use (except cannabis) over the last 3 months, determined by the MINI. Lifetime/present cannabis use (non-disordered levels) will be allowed, given its common usage in individuals in this age range.
13. Current or past psychotic-spectrum disorder
14. History of seizures

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay C Fournier, Ph. D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Transcranial Direct Current Stimulation (tDCS) During fMRI Followed by Active tDCS During fMRI: Each subject will first undergo sham transcranial direct current stimulation while completing a task in the functional magnetic resonance imaging scanner. One week later, they will receive active tDCS during the task in the scanner.
  TDCS - transcranial direct current stimulation: TDCS involves passing a weak current through the brain. One variant, cathodal TDCS, can be used to temporarily hyperpolarize cortical pyramidal cells, thereby decreasing neuronal connections. TDCS has been explored as a possible treatment for depression, but results to date are mixed. No work has examined whether TDCS can be used in an individually guided manner to target locations in the parietal cortex and alter the patterns of circuitry dysfunction described previously.
- ActiveTranscranial Direct Current Stimulation (tDCS) During fMRI Followed by Sham tDCS During fMRI: Each subject will first undergo active transcranial direct current stimulation while completing a task in the functional magnetic resonance imaging scanner. One week later, they will receive sham tDCS during the task in the scanner.
Period: Overall Study
Arm/Group | Sham Transcranial Direct Current Stimulation (tDCS) During fMRI Followed by Active tDCS During fMRI | ActiveTranscranial Direct Current Stimulation (tDCS) During fMRI Followed by Sham tDCS During fMRI
Started | 3 | 1
Completed | 3 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Both Arms Reported Together.: Because only 1 participant entered in the real followed by sham condition, we report baseline variables combined across the arms. All 4 participants received active tDCS.
  TDCS - transcranial direct current stimulation: TDCS involves passing a weak current through the brain. One variant, cathodal TDCS, can be used to temporarily hyperpolarize cortical pyramidal cells, thereby decreasing neuronal connections. TDCS has been explored as a possible treatment for depression, but results to date are mixed. No work has examined whether TDCS can be used in an individually guided manner to target locations in the parietal cortex and alter the patterns of circuitry dysfunction described previously.
Arm/Group | Both Arms Reported Together.
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Quick Inventory Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Range: 0-27. High scores represent more severe depression.
  units on a scale | 11.0 (3.6)
PROMIS Anxiety Short Form [Mean (Standard Deviation); unit: units on a scale] — Range:7-35. Higher scores represent more severe anxiety
  units on a scale | 23.5 (.6)

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level Dependent (BOLD) Response in the Precuneus During an Emotion Regulation Task Completed During fMRI Scanning.
Description: The investigators will determine the effects of TDCS on BOLD response in the precuneus/posterior cingulate gyrus. The BOLD signal is a measure of regional blood flow in the brain and is used as a proxy for neural activity in specific brain regions.
  Values below represent pre-post change in BOLD response to the emotion regulation task that participants complete during fMRI scanning. We hypothesize that tDCS applied to the target used in this study will decrease BOLD signal (lower values) during critical components of this task, normalizing function in this region.
Time Frame: 1 week (between baseline and repeat scanning)
Population: Because no subjects completed the Active followed by Sham tDCS arm, results are reported for the 3 individuals who completed the Sham followed by Active tDCS arm only.
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Active vs Sham Transcranial Direct Current Stimulation During fMRI: Each subject will undergo transcranial direct current stimulation twice while completing a task in the functional magnetic resonance imaging scanner.
  TDCS - transcranial direct current stimulation: TDCS involves passing a weak current through the brain. One variant, cathodal TDCS, can be used to temporarily hyperpolarize cortical pyramidal cells, thereby decreasing neuronal connections. TDCS has been explored as a possible treatment for depression, but results to date are mixed. No work has examined whether TDCS can be used in an individually guided manner to target locations in the parietal cortex and alter the patterns of circuitry dysfunction described previously.
  This is a within subjects design. Each participant received both active and sham treatment in a randomized crossover design. The outcome of interest is the within-person difference in BOLD response between the active and sham tDCS administrations. As such, only one "arm" is reported.
Arm/Group | Active vs Sham Transcranial Direct Current Stimulation During fMRI
Number analyzed (Participants) | 3
arbitrary units | -.09 (.36)

2. Secondary Outcome: The Percentage of Patients Who Reported a Side Effect in the Active tDCS Condition But Not the Sham tDCS Condition
Description: Potential side effects (e.g., headaches, dizziness, uncomfortable sensations, etc...) will be assessed after each tDCS and sham-tDCS administration. Side effects were assessed using a standardized form.
  Count below represents the number of participants who reported a mild or moderate side effect during active tDCS but not sham tDCS.
Time Frame: 30 minutes to 1 hour (the period during which the tDCS device was worn) on each of two scan days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Active vs Sham Transcranial Direct Current Stimulation During fMRI: Each subject will undergo transcranial direct current stimulation twice while completing a task in the functional magnetic resonance imaging scanner.
  TDCS - transcranial direct current stimulation: TDCS involves passing a weak current through the brain. One variant, cathodal TDCS, can be used to temporarily hyperpolarize cortical pyramidal cells, thereby decreasing neuronal connections. TDCS has been explored as a possible treatment for depression, but results to date are mixed. No work has examined whether TDCS can be used in an individually guided manner to target locations in the parietal cortex and alter the patterns of circuitry dysfunction described previously.
  This is a within subjects design. Each participant received both active and sham treatment in a randomized crossover design. The outcome of interest is the number of individuals who reported a side-effect during the active tDCS stimulation but not the sham tDCS stimulation. As such, only one "arm" is reported.
Arm/Group | Active vs Sham Transcranial Direct Current Stimulation During fMRI
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 day (the day of the scan).
Groups:
- Active Transcranial Direct Current Stimulation During fMRI; Sham Transcranial Direct Current Stimulation During fMRI: Each subject will undergo both active and sham transcranial direct current stimulation while completing a task in the functional magnetic resonance imaging scanner.
  TDCS - transcranial direct current stimulation: TDCS involves passing a weak current through the brain. One variant, cathodal TDCS, can be used to temporarily hyperpolarize cortical pyramidal cells, thereby decreasing neuronal connections. TDCS has been explored as a possible treatment for depression, but results to date are mixed. No work has examined whether TDCS can be used in an individually guided manner to target locations in the parietal cortex and alter the patterns of circuitry dysfunction described previously.
  This is a within subjects design. Each participant received both active and sham tDCS in a randomized crossover design. The critical determinant of adverse events due to tDCS is the number reported during the active tDCS condition compared to those reported during the sham tDCS condition. As such, only one "arm" is reported, and it represents the number of events reported during active tDCS that were not reported by the same individual(s) during sham tDCS. 4 cases are reported (rather than 3) out of abundance of caution as one individual received only active tDCS and was lost to follow-up and so could not contribute the necessary data for the primary or secondary outcomes.
Arm/Group | Active Transcranial Direct Current Stimulation During fMRI | Sham Transcranial Direct Current Stimulation During fMRI
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Transcranial Direct Current Stimulation During fMRI (N=4) | Sham Transcranial Direct Current Stimulation During fMRI (N=3)
headache (Nervous system disorders) | 3 (3) | 0 (0)
Scalp burning/itching/tingling sensation (Nervous system disorders) | 4 (4) | 3 (3)
Sleepiness/dizziness (Nervous system disorders) | 3 (3) | 1 (1)
tension/anxiety/disorientation (Nervous system disorders) | 2 (2) | 0 (0) — self-reported increase in tension, anxiety, and/or disorientation
Mood change or difficulty concentrating (Nervous system disorders) | 0 (0) | 2 (2) — Self-reported mood change and/or difficulties concentrating.

LIMITATIONS AND CAVEATS:
This study was closed due to Covid 19 restrictions. Only 3 people completed the protocol. No conclusions should be drawn from the results reported. Because of the low sample size, no statistical analyses were undertaken.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT04598152/Prot_SAP_000.pdf